CLINICAL TRIAL: NCT01152580
Title: Assessing the Efficacy of Melatonin on Bone Health in Peri-menopausal Women
Brief Title: Melatonin Osteoporosis Prevention Study
Acronym: MOPS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duquesne University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 07-88
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Results first posted 2012-03-12 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Osteoporosis; Osteopenia
Keywords: melatonin; menopause; perimenopause; sleep; osteoporosis; osteopenia; anxiety; depression; hypertension
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Anxiety Disorders; Depression; Hypertension | interventions — Melatonin; Sugars; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill (Placebo Comparator)
  Interventions: Dietary Supplement: sugar pill
- melatonin (Active Comparator)
  Interventions: Dietary Supplement: melatonin

INTERVENTIONS:
Dietary Supplement: melatonin — 3mg p.o. at bedtime daily
  Other Names: Nature's Bounty Melatonin; Natrol Melatonin; Spring Valley Melatonin
  Arms: melatonin
Dietary Supplement: sugar pill — lactose p.o. at bedtime daily
  Other Names: Lactose
  Arms: Sugar pill

SUMMARY:
Osteoporosis is one of the most common skeletal disorders. Today in the United States, 10 million individuals have osteoporosis and 34 million more have low bone mass or osteopenia, which places them at an increased risk of some day developing osteoporosis. Of the people affected by this problem, 68% are women.The current thinking on the development of osteoporosis is that the changes in bone turnover that occur with aging play a major factor. Many modalities of treatment are used to prevent the bone loss and increased fracture risk associated with osteoporosis and osteopenia. Melatonin supplementation may be another treatment modality that lowers risk of hip fracture in perimenopausal women. Melatonin can remodel bone in animal models and in culture. Melatonin works through melatonin receptors to form osteoblasts from human mesenchymal stem cells and has been shown to inhibit osteoclast activity in rodents. Melatonin levels have been correlated with modulating bone markers; low nocturnal levels of melatonin correlate with in an increase in bone marker metabolism and osteoporosis. It is been shown that women who have worked night-shifts for greater than 20 years have increased risk for wrist and hip fractures. Night-shift workers have lower nocturnal melatonin levels than people who do not work the night-shift. The addition of exogenous melatonin suppresses bone marker metabolism. In human stem cells taken from bone marrow, melatonin increases the activity of bone-forming cells called osteoblasts. It is hypothesized that melatonin will improve bone health, menopausal quality of life and sleep compared to placebo in perimenopausal women. In particular, the investigators expect perimenopausal women taking melatonin to show an improvement in overall bone health as revealed by a reduction in bone marker turnover since bone resorption increases more so than bone absorption in this population compared to those women taking placebo. We also expect that perimenopausal women taking melatonin to have better control over their menopausal symptoms, better quality of life and less sleep disturbances when compared to their placebo controls since melatonin is known to modulate estrogen levels in the body and regulate sleep. The data from these studies may provide novel and alternative uses for melatonin; in particular its use for the prevention and/or treatment of osteoporosis.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE Osteoporosis is one of the most common skeletal disorders. Today in the United States, 10 million individuals have osteoporosis and 34 million more have low bone mass or osteopenia, which places them at an increased risk of some day developing osteoporosis. Of the people affected by this problem, 68% are women.[1] Osteoporosis is characterized by low bone mass and microarchitectural disruption, such that fewer, thinner bony spicules are present leading to less structural support. These hallmark features of osteoporosis lead to increased skeletal fragility and an increased fracture risk.[2] Hip fracture specifically has been shown to be a major problem leading to increased morbidity and mortality.[3] In addition osteoporotic fractures are responsible for a large portion of health care spending. In 1995 $13.8 billion in health care expenditures were attributable to osteoporotic fractures.[4] Because the health of older adults often deteriorates after hip fracture, efforts to prevent fracture by treating and preventing osteoporosis are critical to reducing this common cause of morbidity, mortality and health service utilization.

The current thinking on the development of osteoporosis is that the changes in bone turnover that occur with aging play a major factor. One study which measured markers of bone formation, such as osteocalcin (OC), and markers of bone resorption, such as type I collagen cross-linked N-telopeptide (NTX), showed that rates of bone formation and resorption are high in elderly women. However, bone resorption increases more so than bone formation leading resorption to be the major determinant of bone mass.[5] These biochemical markers of bone formation and resorption may play an important role in monitoring therapy. In a recent review that examined clinical studies in which bone turnover markers were measured after beginning treatment with a bisphosphonate, the data showed that suppression of bone turnover markers occurred after as little as three months of therapy.[6,7] This suppression in bone turnover markers was also associated with reduction in risk for fracture.[6,7] Although dual X-ray absorptiometry (DXA) is the gold standard for diagnosis of osteoporosis and osteopenia, recent reports are showing that DXA may not be the best method for measuring bone health. For example, bone fractures routinely occur despite modest bone mineral density levels and no significant reduction in the risk of fracture occurs in patients taking one of the two standard medications, one that significantly increases bone mineral density and the other that moderately increases it.[6] Thus, it is currently thought that bone quality may not be clinically assessed by measures other than the determination of bone metabolism with biochemical markers of bone turnover because these markers measure "living" bone cells.[6] Many modalities of treatment are used to prevent the bone loss and increased fracture risk associated with osteoporosis and osteopenia. One method involves use of calcium and vitamin D supplementation such that total calcium intake is approximately 1500 mg/day. Calcium and vitamin D supplementation may increase bone mineral density to a small extent, but not nearly to the same degree as is seen with other treatment modalities.[8] Therefore, it is often combined with another treatment method for better efficacy. Bisphosphonates are being used more and more often in postmenopausal women. These antiresorptive agents have been shown to prevent bone loss and reduce the incidence of vertebral and nonvertebral fractures.[9] Calcitonin has been shown to decrease vertebral fractures, increase bone mineral density at the lumbar spine and inhibit bone turnover.[10]

Melatonin supplementation may be another treatment modality that lowers risk of hip fracture in perimenopausal women. Melatonin can remodel bone in animal models and in culture.[11] Melatonin works through melatonin receptors to form osteoblasts from human mesenchymal stem cells[12] and has been shown to inhibit osteoclast activity in rodents.[13] Melatonin levels have been correlated with modulating bone markers whereby low nocturnal levels of melatonin correlate with in an increase in bone marker metabolism and osteoporosis.[14] The addition of exogenous melatonin suppresses bone marker metabolism.[15] Work from my laboratory reveals that application of melatonin to human bone stem cells grown in culture enhances alkaline phosphatase activity by 50% and calcium deposition by 10-fold.[16]

HYPOTHESIS AND SPECIFIC AIMS We hypothesize that melatonin will improve bone health, menopausal quality of life and sleep compared to placebo in perimenopausal women.

1. Assess the feasibility of recruiting perimenopausal women willing to be enrolled in a randomized, trial of melatonin versus placebo
2. Assess the effects of melatonin versus placebo on markers of bone health, quality of life, and sleep disturbance.

PRIMARY ENDPOINTS: The primary outcome variables are bone turnover marker status, and melatonin levels as measured in blood and bone density as measured by the Achilles method.

SECONDARY ENDPOINTS:

1. Quality of life as measured by the MenQOL, a validated scale of menopausal quality of life
2. Sleep, as measured by the Pittsburgh Sleep Questionnaire

RESEARCH PLAN This study is a longitudinal, cohort trial of 20 subjects who are perimenopausal and aged 45 years old or greater who have new onset of irregular menses not due to other known causes such as polycystic ovaries or hypothyroidism. Perimenopause is defined as the time between the onset of menstrual irregularity and menopause; there is no lab test that is diagnostic of perimenopause. Thus, the investigators will include women who, according to their age, are likely to be perimenopausal (age 45 or greater) and who have symptoms of perimenopause (irregular menses). Once a cohort of 20 subjects is recruited, the investigators will randomize volunteers using a computer-generated blocked randomization scheme. Five study subjects will receive placebo and 15 study subjects will receive melatonin, 3 mg). The women enrolled in the study will be asked to take their treatments by mouth at bedtime each day for 6 months to coincide with the nocturnal surge in melatonin each day. This dose of melatonin has been chosen because 3 mg melatonin is commonly used to induce phase-shifts in circadian rhythms in people.[17] Seeing that this is one of our secondary endpoints, this dose is appropriate. Regarding melatonin's effects on bone, there is nothing known about its efficacy on forming bone in women. Therefore, the dose of melatonin was chosen based on the reported literature using pre-clinical or in vitro culture models that showed positive effects on bone formation. These reports show variable effects of melatonin ranging from 400 pM in rat [15], to 5 mg melatonin in mouse (unpublished data) to 50 nM on human mesenchymal stem cells grown in culture.[12,16] The bioavailability of melatonin is 17% in females taking 250 mcg melatonin po.[18] Thus, a 3 mg dose of melatonin taken by mouth would result in a nocturnal exogenous level of 2.19 mM. The terminal half-life of melatonin is about 41 minutes in females [18], however, accumulation of melatonin in the bone marrow occurs [11]. Therefore, these data suggest that our 3 mg dose is appropriate for these studies.

PLANS FOR ASSESSMENT AND STUDY OUTCOMES Our primary outcome will be the levels of bone turnover markers, OC and NTX, bone density and melatonin taken at baseline and then after 6 months of treatment. The change in bone turnover marker levels will be compared between those taking melatonin and those taking placebo. Baseline levels of OC and NTX will be calculated. For this study the investigators will also visually inspect the data in order to perform descriptive analyses of the demographic characteristics of our population, such as age, and weight. We will explore characteristics of any individuals who have a significant improvement in their bone turnover markers, such as compliance with the treatment, diet, and lifestyle as determined by the diary. We will also make note of characteristics such as current or past cigarette smoking and alcohol and caffeine consumption as individuals with these risk factors may show less improvement in their bone turnover markers. We will use intention to treat as our primary analysis. We will attempt to minimize missing data with careful follow-up of subjects, maintaining consistent contact with them over the study period, and remunerating them for their inconvenience. If a subject drops out of the study, the investigators will still attempt to obtain their follow up studies.

Expected Outcomes.We expect perimenopausal women taking melatonin to show an improvement in overall bone health as revealed by an increase in bone density, an increase in OC and a decrease in NTX levels when compared to those women taking placebo. We also expect those taking melatonin to have better control over their menopausal symptoms, better quality of life and less sleep disturbances compared to their placebo controls. The potential benefits of participating in this study include the possibility of decreasing bone turnover and reducing fracture risk as well as improve sleep regardless, a condition much affected in this population of women. The data from these studies may provide novel and alternative uses for melatonin for the prevention of osteoporosis and provide women with more options to manage diseases associated with menopause.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include perimenopausal women,
* willingness to participate in the 6-month study, willingness to undergo testing of bone turnover markers before and after the drug therapies and willingness to provide a self-assessment on quality of life and sleep throughout the program.
* Subjects must be willing to take their treatments right before bed and to not to consume alcohol with this medication.

Exclusion Criteria:

* Exclusion criteria will include women in whom osteopenia is a result of some other known process such as hyperparathyroidism, metastatic bone disease, multiple myeloma or chronic steroid use.
* Those individuals on osteoporotic drugs, hypnotics, CYP1A2 inhibiting drugs, fluvoxamine or those with severe sleep apnea, severe COPD and those with moderate or severe hepatic impairment will also be excluded.
* Individuals who are lactose intolerant will also be excluded because the placebo and melatonin capsules will contain lactose.

Ages: 45 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2008-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula A Witt-Enderby, PhD, Principal Investigator — Duquesne University School of Pharmacy; Judith L Balk, MD, Principal Investigator — Magee-Womens Hospital, University of Pittsburgh
Locations (1):
- Duquesne University School of Pharmacy Center for Pharmacy Care, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] www.osteo.org. Osteoporosis Overview. National Institute of Health Osteoporosis and Related Bone Disease. June 2005.
- [Background] Parfitt AM, Villanueva AR, Foldes J, Rao DS. Relations between histologic indices of bone formation: implications for the pathogenesis of spinal osteoporosis. J Bone Miner Res. 1995 Mar;10(3):466-73. doi: 10.1002/jbmr.5650100319. PMID 7785469
- [Background] Wolinsky FD, Fitzgerald JF, Stump TE. The effect of hip fracture on mortality, hospitalization, and functional status: a prospective study. Am J Public Health. 1997 Mar;87(3):398-403. doi: 10.2105/ajph.87.3.398. PMID 9096540
- [Background] Ray NF, Chan JK, Thamer M, Melton LJ 3rd. Medical expenditures for the treatment of osteoporotic fractures in the United States in 1995: report from the National Osteoporosis Foundation. J Bone Miner Res. 1997 Jan;12(1):24-35. doi: 10.1359/jbmr.1997.12.1.24. PMID 9240722
- [Background] Garnero P, Sornay-Rendu E, Chapuy MC, Delmas PD. Increased bone turnover in late postmenopausal women is a major determinant of osteoporosis. J Bone Miner Res. 1996 Mar;11(3):337-49. doi: 10.1002/jbmr.5650110307. PMID 8852944
- [Background] Nishizawa Y, Nakamura T, Ohta H, Kushida K, Gorai I, Shiraki M, Fukunaga M, Hosoi T, Miki T, Chaki O, Ichimura S, Nakatsuka K, Miura M; Committee on the Guidelines for the Use of Biochemical Markers of Bone Turnover in Osteoporosis Japan Osteoporosis Society. Guidelines for the use of biochemical markers of bone turnover in osteoporosis (2004). J Bone Miner Metab. 2005;23(2):97-104. doi: 10.1007/s00774-004-0547-6. No abstract available. PMID 15750686
- [Background] Bonnick SL, Shulman L. Monitoring osteoporosis therapy: bone mineral density, bone turnover markers, or both? Am J Med. 2006 Apr;119(4 Suppl 1):S25-31. doi: 10.1016/j.amjmed.2005.12.020. PMID 16563938
- [Background] Riggs BL, O'Fallon WM, Muhs J, O'Connor MK, Kumar R, Melton LJ 3rd. Long-term effects of calcium supplementation on serum parathyroid hormone level, bone turnover, and bone loss in elderly women. J Bone Miner Res. 1998 Feb;13(2):168-74. doi: 10.1359/jbmr.1998.13.2.168. PMID 9495509
- [Background] Hosking D, Chilvers CE, Christiansen C, Ravn P, Wasnich R, Ross P, McClung M, Balske A, Thompson D, Daley M, Yates AJ. Prevention of bone loss with alendronate in postmenopausal women under 60 years of age. Early Postmenopausal Intervention Cohort Study Group. N Engl J Med. 1998 Feb 19;338(8):485-92. doi: 10.1056/NEJM199802193380801. PMID 9443925
- [Background] Chesnut CH 3rd, Silverman S, Andriano K, Genant H, Gimona A, Harris S, Kiel D, LeBoff M, Maricic M, Miller P, Moniz C, Peacock M, Richardson P, Watts N, Baylink D. A randomized trial of nasal spray salmon calcitonin in postmenopausal women with established osteoporosis: the prevent recurrence of osteoporotic fractures study. PROOF Study Group. Am J Med. 2000 Sep;109(4):267-76. doi: 10.1016/s0002-9343(00)00490-3. PMID 10996576
- [Background] Witt-Enderby PA, Radio NM, Doctor JS, Davis VL. Therapeutic treatments potentially mediated by melatonin receptors: potential clinical uses in the prevention of osteoporosis, cancer and as an adjuvant therapy. J Pineal Res. 2006 Nov;41(4):297-305. doi: 10.1111/j.1600-079X.2006.00369.x. PMID 17014686
- [Background] Radio NM, Doctor JS, Witt-Enderby PA. Melatonin enhances alkaline phosphatase activity in differentiating human adult mesenchymal stem cells grown in osteogenic medium via MT2 melatonin receptors and the MEK/ERK (1/2) signaling cascade. J Pineal Res. 2006 May;40(4):332-42. doi: 10.1111/j.1600-079X.2006.00318.x. PMID 16635021
- [Background] Koyama H, Nakade O, Takada Y, Kaku T, Lau KH. Melatonin at pharmacologic doses increases bone mass by suppressing resorption through down-regulation of the RANKL-mediated osteoclast formation and activation. J Bone Miner Res. 2002 Jul;17(7):1219-29. doi: 10.1359/jbmr.2002.17.7.1219. PMID 12096835
- [Background] Ostrowska Z, Kos-Kudla B, Marek B, Kajdaniuk D. Influence of lighting conditions on daily rhythm of bone metabolism in rats and possible involvement of melatonin and other hormones in this process. Endocr Regul. 2003 Sep;37(3):163-74. PMID 14986722
- [Background] Ostrowska Z, Kos-Kudla B, Nowak M, Swietochowska E, Marek B, Gorski J, Kajdaniuk D, Wolkowska K. The relationship between bone metabolism, melatonin and other hormones in sham-operated and pinealectomized rats. Endocr Regul. 2003 Dec;37(4):211-24. PMID 15106818
- [Background] Sethi S, Radio NM, Kotlarczyk MP, Chen CT, Wei YH, Jockers R, Witt-Enderby PA. Determination of the minimal melatonin exposure required to induce osteoblast differentiation from human mesenchymal stem cells and these effects on downstream signaling pathways. J Pineal Res. 2010 Oct;49(3):222-38. doi: 10.1111/j.1600-079X.2010.00784.x. Epub 2010 Jul 6. PMID 20626586
- [Background] Burgess HJ, Revell VL, Eastman CI. A three pulse phase response curve to three milligrams of melatonin in humans. J Physiol. 2008 Jan 15;586(2):639-47. doi: 10.1113/jphysiol.2007.143180. Epub 2007 Nov 15. PMID 18006583
- [Background] Fourtillan JB, Brisson AM, Gobin P, Ingrand I, Decourt JP, Girault J. Bioavailability of melatonin in humans after day-time administration of D(7) melatonin. Biopharm Drug Dispos. 2000 Jan;21(1):15-22. doi: 10.1002/1099-081x(200001)21:13.0.co;2-h. PMID 11038434
- [Result] Kotlarczyk MP, Lassila HC, O'Neil CK, D'Amico F, Enderby LT, Witt-Enderby PA, Balk JL. Melatonin osteoporosis prevention study (MOPS): a randomized, double-blind, placebo-controlled study examining the effects of melatonin on bone health and quality of life in perimenopausal women. J Pineal Res. 2012 May;52(4):414-26. doi: 10.1111/j.1600-079X.2011.00956.x. Epub 2012 Jan 6. PMID 22220591
- See also: Osteoporosis Overview. National Institute of Health Osteoporosis and Related Bone Disease. June 2005 — http://www.osteo.org
- See also: Melatonin Osteoporosis Prevention Study (MOPS): A Randomized, Double-Blind, Placebo-Controlled Study Examining the Effects of Melatonin on Bone Health and Quality of Life in Perimenopausal Women — http://www.ncbi.nlm.nih.gov/pubmed/22220591

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in September, 2008 and continued through February, 2010 using neighborhood and city newspapers, posting of flyers, on-campus advertising and news features in campus, local and city newspapers and the local news. Eligible subjects reported to the Center for Pharmacy Care at Duquesne University for screenings and assessments.
Pre-assignment Details: Eligible subjects were randomly assigned using a computer-generated randomization scheme to receive either placebo or melatonin at a 3:1 ratio (treatment:placebo). Participants and principle investigators were completely blinded to the group assignments throughout the entire study thus achieving allocation concealment.
Groups:
- Sugar Pill: Each capsule contained lactose and the study subjects took this nightly, p.o. for 6 months
- Melatonin: Each capsule contained 3 mg melatonin and each subject was asked to take this nightly p.o. for 6 months
Period: Overall Study
Arm/Group | Sugar Pill | Melatonin
Started | 5 | 14
Completed | 5 | 13
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Melatonin | Total
Number analyzed (Participants) | 5 | 13 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 13 | 18
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47.5 (2.0) | 50.3 (3) | 49.5 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 18
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 13 | 18
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 13 | 18
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 21.7 (3.5) | 25.7 (3.7) | 24.6 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Melatonin (3 mg) or Placebo on the Mean Change in Serum Osteocalcin (OC) Levels in Women After 6 Months, as Compared to Baseline
Description: Osteocalcin is a measure of osteoblast activity because it is secreted from osteoblasts. Osteocalcin levels were measured in the serum of women at baseline and after 6 months of taking placebo or melatonin (3 mg) and the data are reported as ng/mL. Osteoblasts are bone-forming cells so a more positive mean change in osteoblast activity over time (6 months - baseline) could indicate an improvement in bone mineral density. A more negative mean change in osteocalcin levels over time (6 months - baseline) could indicate a worsening of bone mineral density.
Time Frame: Baseline and 6 months
Population: intention to treat
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sugar Pill | Melatonin
Number analyzed (Participants) | 5 | 13
ng/mL | -0.6 (0.596) | 1.83 (1.066)

2. Secondary Outcome: The Effect of Melatonin (3 mg) or Placebo on the Mean Change in Menopause-Specific Quality of Life (MENQOL) Physical Domain Scores in Women After 6 Months, as Compared to Baseline.
Description: Menopause-Specific Quality of Life (MENQOL) questionnaires were administered to women at baseline and after 6 months of taking placebo or melatonin nightly. The MENQOL is a validated questionnaire that measures 4 domains of menopause quality of life in women: physical, vasomotor, psychosocial and sexual with each domain having a scale of "not bothered" (score 0) or "bothered ranging from 1(not too bothered) to 6 (really bothered)". A more negative mean change for each of the MENQOL domain scores indicates an improvement of these symptoms and a more positive value a worsening of symptoms.
Time Frame: Baseline and 6 mos
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Melatonin
Number analyzed (Participants) | 5 | 13
units on a scale | 0.1 (0.5) | -0.6 (0.8)

3. Secondary Outcome: The Effect of Melatonin (3 mg) or Placebo on the Mean Change in Menopause-Specific Quality of Life (MENQOL) Vasomotor Domain Scores in Women After 6 Months, as Compared to Baseline.
Description: as for outcome 2
Time Frame: Baseline and 6 mos
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Melatonin
Number analyzed (Participants) | 5 | 13
units on a scale | -0.2 (0.4) | 0.4 (1.8)

4. Primary Outcome: The Effect of Melatonin (3 mg) or Placebo on the Mean Change in Serum Type-1 Collagen Cross-linked N-telopeptide (NTX) Levels in Women After 6 Months, as Compared to Baseline.
Description: Type-1 collagen cross-linked N-telopeptide (NTX) levels were measured in the serum of women at baseline and after taking placebo or melatonin (3 mg) nightly for 6 months. NTX, reported as bone collagen equivalents (BCE), is released from bone due to the actions of osteoclasts or bone breakdown cells. A more positive mean change in NTX levels (6 months - baseline) could result in a worsening of bone mineral density due to an increase in bone breakdown whereas a more negative mean change in NTX levels could result in an improvement in bone mineral density due to a decrease in bone breakdown.
Time Frame: Baseline and 6 months
Population: intention to treat
Measure: Mean (Standard Deviation); unit: nM BCE
Arm/Group | Sugar Pill | Melatonin
Number analyzed (Participants) | 5 | 13
nM BCE | -0.36 (0.97) | -0.32 (1.4)

5. Secondary Outcome: The Effect of Melatonin (3 mg) or Placebo on the Mean Change in Menopause-Specific Quality of Life (MENQOL) Psychosocial Domain Scores in Women After 6 Months, as Compared to Baseline.
Description: as for outcome 2
Time Frame: Baseline and 6 mos
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Melatonin
Number analyzed (Participants) | 5 | 13
units on a scale | -0.2 (1.3) | -0.4 (1.3)

6. Primary Outcome: The Effect of Melatonin (3 mg) or Placebo on the Mean Change in Bone Density in Women After 6 Months, as Compared to Baseline.
Description: The mean change in bone mineral density (BMD), represented by T-scores, was assessed by calcaneal ultrasound in women taking melatonin (3 mg) or placebo nightly at baseline and after 6 months. A T-score is a comparison of a subject's BMD to that of a healthy 30 year old female of the same ethnicity. The more negative the T-score, the worse the BMD. Osteoporosis or brittle bone disease is defined as a T-score -2.5 or less. A more negative mean change in a T-score would indicate a worsening of BMD. A more positive mean change in a T-score would indicate an improvement of BMD.
Time Frame: Baseline and 6 months
Population: intention to treat
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Sugar Pill | Melatonin
Number analyzed (Participants) | 5 | 13
T-score | -0.02 (0.113) | 0.05 (0.01)

7. Secondary Outcome: The Effect of Melatonin (3 mg) or Placebo on the Mean Change in Menopause-Specific Quality of Life (MENQOL) Sexual Domain Scores in Women After 6 Months, as Compared to Baseline.
Description: as for outcome 2
Time Frame: Baseline and 6 mos
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Melatonin
Number analyzed (Participants) | 5 | 13
units on a scale | -0.7 (1.4) | -0.4 (1.2)

8. Secondary Outcome: The Effect of Melatonin (3 mg) or Placebo on the Mean Change in the Pittsburgh Sleep Quality Index (PSQI) in Women After 6 Months, as Compared to Baseline.
Description: Pittsburgh Sleep Quality Index (PSQI) Questionnaire is a validated questionnaire that assesses the quality and quantity of sleep and sleep disorders.This survey is designed to identify "good" and "poor" sleepers and has a score scale that ranges from "0-21" with "0" being good quality of sleep and "21" being poor quality of sleep and/or indicating as having a sleep disorder. A more positive mean change in the PSQI over time indicates a worsening of sleep. A more negative mean change in the PSQI over time indicates an improvement in sleep.
Time Frame: Baseline and 6 months
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Melatonin
Number analyzed (Participants) | 5 | 13
units on a scale | -1.0 (1.4) | -0.5 (2.8)

ADVERSE EVENTS:
Arm/Group | Sugar Pill | Melatonin
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/13
Other Adverse Events (participants affected / at risk) | 0/5 | 0/13

LIMITATIONS AND CAVEATS:
Limitations to this study include small sample sizes, length of follow-up, and heterogeneity in terms of stage of perimenopause and prevalence of menopausal symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No